CLINICAL TRIAL: NCT01774448
Title: The Efficacy of Mindfulness-Based Cognitive Therapy (MBCT) to Improve Depression Symptoms and Quality of Life in Individuals With Dementia and Their Caregivers: A Pilot Study
Brief Title: Mindfulness Research Program: Designed to Enhance Wellbeing in People Living With Dementia and Their Spouses
Acronym: MBCT_AD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lakehead University (Other)
Collaborators: Alzheimer Society of Canada (Other)
Responsible Party: Principal Investigator, Michel Bédard, Full Professor, Lakehead University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: ASC-1309
Record Dates: First submitted 2013-01-14; First posted 2013-01-24 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Dementia
Keywords: Dementia; Spouse Caregiver; Depression; Mind Body Therapy; Cognitive Therapy; Quality of Life; Attention; Memory
MeSH Terms: conditions — Dementia; Depression | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Waitlist Control (No Intervention): Participants in the control group will undergo a non-intervention 8-week period while on the 'waitlist control' then will be crossed-over to the Mindfulness-Based Cognitive Therapy intervention.
- Mindfulness-Based Cognitive Therapy (Experimental): Mindfulness-Based Cognitive Therapy is an 8-week intervention, one session per week for 2 hours, where participants will learn and practice formal and informal mindfulness meditation, and participate in group discussion and inquiry.
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy

INTERVENTIONS:
Behavioral: Mindfulness-Based Cognitive Therapy — In the experimental condition, individuals with dementia (n = 15) and their spouses (n = 15) will partake in one MBCT session per week for 8 weeks. The partners will attend separate MBCT sessions (different day of the week). In the control condition, individuals with dementia (n = 15) and their spouses (n= 15) will go through an 8-week waitlist control period.
  Arms: Mindfulness-Based Cognitive Therapy

SUMMARY:
People with dementia forget things and have trouble concentrating. In addition, they and their caregivers can become depressed. This project will show whether Mindfulness-Based Cognitive Therapy (MBCT) can lessen depression, increase attention spans and improve quality of life for those affected by the disease and their caregivers.

MBCT combines intensive training in mindfulness meditation with Cognitive Behavioural Therapy. Studies show the meditation component creates changes in areas of the brain associated with our ability to pay attention. This form of meditation can help those impacted by dementia become more aware of their depressive thinking, leading to improved ways of coping.

The investigators predict that individuals in the early stages of dementia and their spousal caregivers will report fewer depression symptoms following the 8-week Mindfulness-Based Cognitive Therapy (MBCT) Program, as well as experience improvements in quality of life and daily mindfulness.

If successful, MBCT could improve the quality of life in individuals with dementia and their caregivers, as well as may take pressure off the health care system by delaying institutionalization.

DETAILED DESCRIPTION:
The overall objective of the proposed study is to investigate the efficacy of Mindfulness-Based Cognitive Therapy (MBCT) to alleviate depression symptoms, increase attention abilities, and improve quality of life in individuals with dementia and their caregivers. MBCT works to help individuals increase concentration and increase awareness of depressive thinking to ultimately provide a better means of coping and emotional regulation.

While dementia is non-reversible and progressive in nature, supportive interventions, especially at the early stage of the disease, can make life more manageable for both dementia individuals and their caregivers. Along with the initial signs of forgetfulness and concentration difficulties, it is common for both individuals with dementia and their primary caregivers to also experience depression symptoms. For dementia individuals, depression symptoms are common early on as they still have insight into their disease. This increase in depression has been shown to be related to apathy, overall poorer quality of life and cognitive decline. Caregivers not only witness a significant change in daily functioning of someone they love and know well, they are also faced with new responsibilities associated with managing the disease, while simultaneously trying to juggling their own day-to-day tasks. These drastic changes and increased responsibilities have been shown to increase feelings of depression and burden, resulting in coping-related problems in caregivers.

Counseling intervention in early stages of dementia has been shown to delay and even decrease patient admittance into long-term facilities, ultimately relieving stress placed on the healthcare system. MBCT is a specific program designed to, and proven successful at, treating various populations with recurrent depression. With its unique therapeutic approach of integrating intensive training in mindfulness meditation with Cognitive Behavioural Therapy, MBCT helps individuals pay greater attention, increase concentration, increase awareness of depressive thinking and learn to apply more skillful means of coping. In addition to treating depression, the meditation component of MBCT has also been shown to improve various aspects of attention and result in changes in neural networks implicated in attention processes. The investigators predict that MBCT will alleviate depression symptoms and increase quality of life in both patients and caregivers. The investigators also expect that individuals will experience improvements in attention and memory abilities.

If successful, MBCT could improve overall quality of life in dementia individuals and caregivers, as well as benefit our healthcare system by delaying institutionalization. From a research perspective, success of this program may lead to a larger clinical controlled trial to further investigate the efficacy of MBCT in individuals affected by dementia.

ELIGIBILITY:
Inclusion Criteria:

* Early stages of dementia
* Spousal caregiver (no signs of dementia/mild cognitive impairment)
* Evidence of at least mild depression (in at least one partner)
* Speak, read, and write in English

Exclusion Criteria:

* Neurological Disorder (other than dementia for dementia group)
* Psychological Disorder

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in Depression Symptoms | 10 weeks
  Change score on Geriatric Depression Scale: Change from pre-intervention baseline depression symptoms (Week 1) at post-intervention (Week 10).

SECONDARY OUTCOMES:
Change in Apathy Levels | 10 weeks
  Change score on Apathy Evaluation Scale: Change from pre-intervention baseline apathy levels (Week 1) at post-intervention (Week 10).
Change in Quality of Life | 10 weeks
  Change score on Quality of Life-AD Scale: Change from pre-intervention baseline quality of life (Week 1) at post-intervention (Week 10).
Change in Anxiety Levels | 10 weeks
  Change score on Depression, Anxiety and Stress Scale: Change from pre-intervention baseline anxiety symptoms (Week 1) at post-intervention (Week 10).
Change in Levels of Coping | 10 Weeks
  Change score on the Brief COPE: Change from pre-intervention baseline levels of coping (Week 1) at post-intervention (Week 10).
Change in Burden Levels | 10 Weeks
  Change score on Zarit Burden Inventory: Change from pre-intervention baseline burden levels (Week 1) at post-intervention (Week 10).
Change in Levels of Self-Compassion | 10 weeks
  Change score on Self-Compassion Scale: Change from pre-intervention baseline level of self-compassion (Week 1) at post-intervention (Week 10).
Change in Cognitive Functioning | 10 Weeks
  Change score on Montreal Cognitive Assessment (MoCA): Change from pre-intervention baseline cognitive functioning (Week 1) at post-intervention (Week 10).
Change in Cognitive Functioning | 10 weeks
  Change score on Modified Mini-Mental State Exam (3MS): Change from pre-intervention baseline cognitive functioning (Week 1) at post-intervention (Week 10).
Change in Working Memory | 10 Weeks
  Change score on Digit Span Forward and Backward: Change from pre-intervention baseline working memory (Week 1) at post-intervention (Week 10).
Change in Cognitive Flexibility | 10 weeks
  Change score on Trail Making A and B Tasks: Change from pre-intervention baseline cognitive flexibility (Week 1) at post-intervention (Week 10).
Change in Verbal Fluency | 10 weeks
  Change score on Category Fluency Test: Change from pre-intervention baseline verbal fluency (Week 1) at post-intervention (Week 10).
Change in Short-Term Verbal Memory | 10 weeks
  Change score on trial one of California Verbal Learning Test: Change from pre-intervention baseline verbal memory (Week 1) at post-intervention (Week 10).
Change in Attention | 10 weeks
  Change score on Attention Network Task: Change from pre-intervention baseline attention (Week 1) at post-intervention (Week 10).
Change in Depression Symptoms | 10 weeks
  Change score on Depression, Anxiety, and Stress Scale: Change from pre-intervention baseline depression symptoms (Week 1) at post-intervention (Week 10).
Change in Levels of Mindfulness | 10 weeks
  Change score on 5 Facet Questionnaire: Change from pre-intervention baseline mindfulness levels (Week 1) at post-intervention (Week 10).

CONTACTS AND LOCATIONS:
Overall Officials: Lana J Ozen, PhD, Principal Investigator — Lakehead University; Michel Bedard, PhD, Study Director — Lakehead University